CLINICAL TRIAL: NCT03794869
Title: Short-term Effects of Exercise Program Versus Electropuncture on Pain, Depression, Range of Motion and Disability, in Patients With Chronic Non-specific Low Back Pain: A Randomized Clinical Trial.
Brief Title: Short-term Effects of Exercise Program Versus Electropuncture in Patients With Chronic Non-specific Low Back Pain: A Randomized Clinical Trial.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Almeria (Other)
Responsible Party: Principal Investigator, Adelaida María Castro-Sánchez, PhD(Lecturer), Universidad de Almeria
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UAL-477
Record Dates: First submitted 2019-01-03; First posted 2019-01-07 (Actual); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Low Back Pain; Exercise Program; Electroacupuncture
Keywords: chronic low back pain; physical therapy; randomized clinical trial; exercise program
MeSH Terms: conditions — Low Back Pain | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Single-Blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise program (Experimental): It will be consist in a program of lumbo-pelvic stabilization exercises and strengthening of the core: awareness of breathing, front and side plate abdominal, glute bridge/hip elevations, lift extended leg, pelvic tilt, hamstring stretch, strengthening lower abdominals, cat-camel posture, trunk rotations with flexed knees, rolling in sitting and lumbar extension with hip extensión in prone
  Interventions: Other: Percutaneous electrostimulation treatment (EPS)
- Percutaneous electrostimulation treatment (EPS) (Active Comparator): Apply dry needles in a tight band of some of the muscles that most affect the appearance of low back pain, such as: paravertebral, lumbar quadrate, gluteus medius and pyramidal, and administer analgesic microcurrents.
  Interventions: Other: Exercise program

INTERVENTIONS:
Other: Percutaneous electrostimulation treatment (EPS) — Apply dry needles in a tight band of some of the muscles that most affect the appearance of low back pain, such as: paravertebral, lumbar quadrate, gluteus medius and pyramidal, and administer analgesic microcurrents.
  Arms: Exercise program
Other: Exercise program — It will be consist in a program of lumbo-pelvic stabilization exercises and strengthening of CORE.
  Arms: Percutaneous electrostimulation treatment (EPS)

SUMMARY:
This study evaluate the effectiveness that exists when performing a treatment based on a table of exercises for strengthening the lumbar muscles versus a treatment based on electropuncture in patients with chronic low back pain.

DETAILED DESCRIPTION:
Low back pain has a high prevalence in all European countries, appearing as the main cause of activity limitation in people under 45 years of age. It has got a high recurrence, which decreases the activities of daily life, facilitates the focus of attention to pain and increases the fear of movement, with the consequent muscular atrophy. A serie cases will be conducted comparing a a table of exercises versus electropuncture.

Objective: Evaluate the effectiveness that exists when performing a tratment based on a table of exercises for strengthening the lumbar muscles versus a treatment based on electropuncture.

Methods: A sample of 12 subjects with chronic low back pain will be assigned to an exercise program or dry electropuncture treatment (EPS), during 4 weeks (2 sessions/week). The measurement variables selected for the study were the followings: Straight Leg Raise, Vasalva, Gaesslen test, algometry (pressure pain threshold), goniometry (measurement of the range of motion), Scale of disability for low back pain of Oswestry, Beck's Depression Inventory (BDI), Visual Analogue Scale (EVA), Mcquade's Test and the Roland-Morrys' Questionnaire, developing a pre-treatment and post-treatment assessment.

ELIGIBILITY:
Inclusion Criteria:

* Chronic non-specific low back pain persisting ≥ 3 months.
* Age between 25 and 60 years.
* Not currently receiving physical therapy.

Exclusion Criteria:

* Presence of lumbar stenosis.
* Presence of clinical signs of radiculopathy.
* Diagnosis of spondylolisthesis.
* Diagnosis of fibromyalgia.
* Treatment with corticosteroid or pharmachological medication within the paset 2 weeks.
* A history of spinal surgery.
* Central or peripheral nervous system disease

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2018-04-15 (Actual); Primary Completion 2018-04-16 (Actual); Study Completion 2018-05-16 (Actual)

PRIMARY OUTCOMES:
Algometry | At baseline and immediate post-treatment
  An instrument for measuring the degree of sensitivity to pain.

SECONDARY OUTCOMES:
Goniometry | At baseline and immediate post-treatment
  Measurement of the range of motion
Beck's Depression Inventory | At baseline and immediate post-treatment
  The state of depression will be determined with the Beck Depression Inventory (BDI), a self-applied 21-item questionnaire that assesses a wide spectrum of depressive symptoms. It focuses on the cognitive components of depression, which represent around 50% of the total questionnaire score.
Visual Analog Scale | At baseline and immediate post-treatment
  Pain will be assessed with the Visual Analog Scale (VAS), which assesses the pain intensity and degree of relief experienced by the patient (scored of 0 = no pain; 10 = unbearable pain).
Oswestry Low Back Pain Disability Index. | At baseline and immediate post-treatment
  It has 10 items associated to activities of daily living, each item has a puntuation fron 0 to 5 points
Roland-Morrys' Questionnaire | At baseline and immediate post-treatment
  This is a self-reported questionnaire consisting in 24 items reflecting limitations in different activities of daily living attributed to low back pain including walking, vending over, sitting, lying down, dressing, sleeping, self-care and daily activities
Mcquade Test | At baseline and immediate post-treatment
  It measures the isometric endurance of trunk flexion muscles

CONTACTS AND LOCATIONS:
Locations (1):
- Almeria University, Almería, Spain

REFERENCES:
- [Background] Haas M, Groupp E, Kraemer DF. Dose-response for chiropractic care of chronic low back pain. Spine J. 2004 Sep-Oct;4(5):574-83. doi: 10.1016/j.spinee.2004.02.008. PMID 15363431
- [Background] Pérez Guisado J. Contribución al estudio de la lumbalgia inespecífica. Rev Cubana Ortop Traumatol. 2006;20(2).
- [Background] Hernandez GA, Zamora Salas JD. [Exercise as a treatment for low back pain management]. Rev Salud Publica (Bogota). 2017 Jan-Feb;19(1):123-128. doi: 10.15446/rsap.v19n1.61910. Spanish. PMID 30137166
- [Background] Sekendiz B, Cug M, Korkusuz F. Effects of Swiss-ball core strength training on strength, endurance, flexibility, and balance in sedentary women. J Strength Cond Res. 2010 Nov;24(11):3032-40. doi: 10.1519/JSC.0b013e3181d82e70. PMID 20940644
- [Background] Castro-Sanchez AM, Lara-Palomo IC, Mataran-Penarrocha GA, Fernandez-Sanchez M, Sanchez-Labraca N, Arroyo-Morales M. Kinesio Taping reduces disability and pain slightly in chronic non-specific low back pain: a randomised trial. J Physiother. 2012;58(2):89-95. doi: 10.1016/S1836-9553(12)70088-7. PMID 22613238
- [Background] Meucci RD, Fassa AG, Faria NM. Prevalence of chronic low back pain: systematic review. Rev Saude Publica. 2015;49:1. doi: 10.1590/S0034-8910.2015049005874. Epub 2015 Oct 20. PMID 26487293
- [Background] Lizier DT, Pérez V, Sakata K. Ejercicios para el tratamiento de la lumbálgia inespecífica. Rev. Bras. Anestesiol. 2012;62(6):842-846.
- [Background] Mehrparvar AH, Heydari M, Mirmohammadi SJ, Mostaghaci M, Davari MH, Taheri M. Ergonomic intervention, workplace exercises and musculoskeletal complaints: a comparative study. Med J Islam Repub Iran. 2014 Jul 16;28:69. eCollection 2014. PMID 25405134
- [Background] Goldby LJ, Moore AP, Doust J, Trew ME. A randomized controlled trial investigating the efficiency of musculoskeletal physiotherapy on chronic low back disorder. Spine (Phila Pa 1976). 2006 May 1;31(10):1083-93. doi: 10.1097/01.brs.0000216464.37504.64. PMID 16648741
- [Background] Slade SC, Keating JL. Trunk-strengthening exercises for chronic low back pain: a systematic review. J Manipulative Physiol Ther. 2006 Feb;29(2):163-73. doi: 10.1016/j.jmpt.2005.12.011. PMID 16461178
- [Background] Slade SC, Keating JL. Unloaded movement facilitation exercise compared to no exercise or alternative therapy on outcomes for people with nonspecific chronic low back pain: a systematic review. J Manipulative Physiol Ther. 2007 May;30(4):301-11. doi: 10.1016/j.jmpt.2007.03.010. PMID 17509439
- [Background] Angel Garcia D, Martinez Nicolas I, Saturno Hernandez PJ, Lopez Soriano F. [Clinical approach to chronic lumbar pain: a systematic review of recommendations included in existing practice guidelines]. An Sist Sanit Navar. 2015 Jan-Apr;38(1):117-30. doi: 10.23938/ASSN.0059. Spanish. PMID 25963464
- [Background] Barlas P, Ting SL, Chesterton LS, Jones PW, Sim J. Effects of intensity of electroacupuncture upon experimental pain in healthy human volunteers: a randomized, double-blind, placebo-controlled study. Pain. 2006 May;122(1-2):81-9. doi: 10.1016/j.pain.2006.01.012. Epub 2006 Mar 9. PMID 16527396
- [Background] Mayor D. Electroacupunture: a practical manual and resource. Churchill Livingstone, 2007.
- [Background] Hamza MA, Ghoname EA, White PF, Craig WF, Ahmed HE, Gajraj NM, Vakharia AS, Noe CE. Effect of the duration of electrical stimulation on the analgesic response in patients with low back pain. Anesthesiology. 1999 Dec;91(6):1622-7. doi: 10.1097/00000542-199912000-00012. PMID 10598602
- [Background] Tsukayama H, Yamashita H, Amagai H, Tanno Y. Randomised controlled trial comparing the effectiveness of electroacupuncture and TENS for low back pain: a preliminary study for a pragmatic trial. Acupunct Med. 2002 Dec;20(4):175-80. doi: 10.1136/aim.20.4.175. PMID 12512791
- [Background] Baldry PE. Acupunture, trigger points and musculoeskeletal pain, 2ª ed. London: Churchill Livingstone;1993.
- [Background] Arroyo Fernández R, Martón Villalvilla R, Baldán Bernardino N, Mayoral del Moral O, Salvat Salvat I. Fisioterapia invasiva del síndrome de dolor miofascial: manual de punción seca de puntos gatillos. Panamericana; 2017.
- [Background] Sanabria AM. Prevalencia de dolor lumbar y su relación con factores de riesgo biomecánicos en personal de enfermería. 2015;37(4):319-330.
- [Background] Vera-García F. Core stability: evaluación y criterios para su entrenamiento. Rev. Andaluza de Medicina del Deporte. 2015;(8(3):130-137.
- [Background] Waddell G, Newton M, Henderson I, Somerville D, Main CJ. A Fear-Avoidance Beliefs Questionnaire (FABQ) and the role of fear-avoidance beliefs in chronic low back pain and disability. Pain. 1993 Feb;52(2):157-168. doi: 10.1016/0304-3959(93)90127-B. PMID 8455963
- [Background] Piovesan EJ, Tatsui CE, Kowacs PA, Lange MC, Pacheco C, Werneck LC. [Using algometry of pressure measuring the threshold of trigeminal pain perception in normal volunteers: a new protocol of studies]. Arq Neuropsiquiatr. 2001 Mar;59(1):92-6. doi: 10.1590/s0004-282x2001000100019. French. PMID 11299439
- [Background] Martín S, Arroyo R, Baldán N, Martín T, Mayoral O. Electroestimulación percutánea del punto gatillo miofascial: efectos de la frecuencia sobre el umbral de dolor a la presión. Cuest Fisioter. 2014;43(2):110-120.
- [Background] Manning DC, Rowlingson JC. Back pain and the role of neural blockade. Neural blockade in clinical anesthesia and management of pain. 3º ed. Philadelphia 1998;879.
- [Background] Medrano García R, Varela Hernández A, de la Torre Rosés M, Mendoza Cisneros R. Propuesta de modificación del algoritmo europeo de manejo de la lumbalgia inespecífica. 2010;14(4).